CLINICAL TRIAL: NCT04465058
Title: Clinical Characteristics and Outcome in Critically Ill COVID 19 Patients
Brief Title: Characteristics of Critically Ill COVID 19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hamed, lecturer of anaesthesia, Assiut University
Other Study IDs: yte
Record Dates: First submitted 2020-07-08; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: COVID19 — viral infection

SUMMARY:
COVID19 is n outbreak with unpredictable outcome

ELIGIBILITY:
Inclusion Criteria:

* COVID 19 patients need oxygen therapy

Exclusion Criteria:

* patients does not need oxygen therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: crirical patients need oxygen therapy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2020-08-08 (Estimated); Study Completion 2020-08-10 (Estimated)

PRIMARY OUTCOMES:
clinical characteristics | 48 hours
  measurements of arterial blood gas

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt